CLINICAL TRIAL: NCT01182324
Title: The PTC124 (Ataluren) Clinical Trial for Duchenne Muscular Dystrophy: Exploration of the Experiences of Parents, Clinician Researchers, and the Industry Sponsor
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910171; 10-HG-N171
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-06-24

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Expectations; Duchenne Muscular Dystrophy; Clinical Trial; Motivations
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to describe the experiences of parents, clinician researchers, and industry professionals who were involved in phase II clinical trials of Ataluren for Duchenne muscular dystrophy. We are especially interested in learning about motivations for being involved in the clinical trial, expectations of the trial, the experience of the trial, and relationships between the parents of children involved in the trial, the clinician researchers, and PTC Therapeutics. In addition, we would like to learn more about whether and how families and advocacy organizations experiences in following the progress of the drug, encouraging the clinical trial, and supporting the phase II trials may have affected participants thoughts and feelings about the study.

DETAILED DESCRIPTION:
Some aspects of the traditional process for the development of new potential therapeutics for rare disorders and the ensuing research on safety and efficacy are changing. This is due, in part, to the increased ability of families, parents, individuals with rare disorders, and advocacy organizations to access and control information, to provide monetary or other incentives, and to communicate directly with biopharmaceutical companies and clinical investigators. Increasingly, advocacy organizations (and by extension, the families they serve) create or participate in disorder registries intended to facilitate research by industry and access of families to clinical trials; fund promising bench and clinical research; and lobby for outcomes beneficial to drug developers and researchers, such as increased funding or facilitated FDA approval. The involvement of families in the research process is likely to have implications for how willing individuals are to participate in studies, their expectations and perceptions of the study experience, and their behavior during the study. Their increased level of involvement may also affect how families perceive and respond to a clinical trial in which the results are not as promising as hoped, as quickly as hoped. This partnership approach has implications for biopharmaceutical companies who sponsor treatment trials and for clinical investigators who lead and implement the trials. This qualitative interview study aims to describe, from the perspectives of parents of children involved in a clinical trial, research clinicians implementing the trial, and the company sponsoring the trial, the experience of this new, more collaborative research process. In this case, we will examine the Ataluren trial for Duchenne muscular dystrophy. The results from this study are hypothesis-generating for downstream research and can inform biopharmaceutical companies and clinician researchers as they plan and implement clinical trials for rare disorders and help guide advocacy groups and parent advocates as they partner with researchers and industry.

ELIGIBILITY:
* INCLUSION CRITERIA:
* US residents over 18 years of age who have at least one child with Duchenne Muscular Dystrophy who was enrolled in the phase IIa extension trial or phase IIb trial of PTC124. Participants must be a primary caregiver for their children, must have been involved in deciding whether the child would participate in the clinical trial, and must have accompanied their child to at least one visit to the clinical trial site.
* Clinician researchers over 18 years of age who were involved with implementing the clinical trial at a study site.
* Representatives of PTC Therapeutics over 18 years of age.

All participants must be willing and able to complete an approximately 1-hour long telephone interview in English.

EXCLUSION CRITERIA:

-Must meet inclusion criteria.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07-30; Study Completion 2013-06-24

PRIMARY OUTCOMES:
To describe, inclusive of the perspectives and voices of all of the major participants, the shared experiences of parents, clinician researchers, and industry professionals who were involved in phase II clinical trials for Duchenne Muscular Dyst...

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cohen PD, Herman L, Jedlinski S, Willocks P, Wittekind P. Ethical issues in clinical neuroscience research: a patient's perspective. Neurotherapeutics. 2007 Jul;4(3):537-44. doi: 10.1016/j.nurt.2007.04.008. PMID 17599719
- [Background] Holroyd J, Guthrie D. Family stress with chronic childhood illness: cystic fibrosis, neuromuscular disease, and renal disease. J Clin Psychol. 1986 Jul;42(4):552-61. doi: 10.1002/1097-4679(198607)42:43.0.co;2-8. PMID 3745452
- [Background] Webb CL. Parents' perspectives on coping with Duchenne muscular dystrophy. Child Care Health Dev. 2005 Jul;31(4):385-96. doi: 10.1111/j.1365-2214.2005.00518.x. PMID 15948875